CLINICAL TRIAL: NCT00004909
Title: The Impact of Oral Chemotherapy on Quality of Life in Patients With Recurrent Epithelial Ovarian Cancer
Brief Title: Effect of Chemotherapy Given Either by Mouth or by Infusion on the Quality of Life of Patients With Recurrent Ovarian Epithelial Cancer
Status: Completed | Type: Observational
Sponsor: Northwestern University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Elizabeth Calhoun, Northwestern University
Other Study IDs: NU 98Q3; NU-98Q3; NCI-G00-1694
Record Dates: First submitted 2000-03-07; First posted 2004-03-16 (Estimated); Last update posted 2011-02-21 (Estimated); Status verified 2011-02

CONDITIONS: Ovarian Cancer; Malignant Tumor of Peritoneum; Quality of Life
Keywords: recurrent ovarian epithelial cancer; peritoneal cavity cancer; quality of life
MeSH Terms: conditions — Ovarian Neoplasms; Carcinoma, Ovarian Epithelial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Oral chemotherapy
- Parenteral chemotherapy

SUMMARY:
RATIONALE: Quality-of-life assessment in patients undergoing cancer treatment may help determine the intermediate- and long-term effects of the treatment on these patients.

PURPOSE: This clinical trial studies the effects of chemotherapy given by mouth versus chemotherapy given by infusion on quality of life in patients with recurrent ovarian epithelial cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the impact of oral versus parenteral chemotherapy on quality of life (QOL) in patients with recurrent ovarian epithelial cancer. II. Evaluate the QOL over time in this patient population. III. Determine the impact of disease symptoms, treatment side effects, performance status, and CA-125 levels on QOL assessment in this patient population.

OUTLINE: Patients receive a baseline quality of life (QOL) assessment, an attitudes/preference survey, and a performance status assessment at the time of diagnosis of recurrent disease. Patients are nonrandomly assigned to treatment with either IV or oral chemotherapy using drugs based on National Comprehensive Cancer Network guidelines, prior treatment history, and patient preference. QOL and performance status assessments are obtained again at 3 and 6 months during treatment. Attitudes/preferences are assessed at 6 months. Patients are withdrawn from study if treatment regimen is changed from oral to IV, or from IV to oral during this 6 months.

PROJECTED ACCRUAL: A total of 74 patients will be accrued for this study over 12 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Newly diagnosed recurrent ovarian epithelial cancer or recurrent primary peritoneal cancer as evidenced by new clinical or radiologic detected mass or rising serum CA-125 level No progressive disease with ongoing treatment

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: Not specified Life expectancy: Not specified Hematopoietic: Not specified Hepatic: Not specified Renal: Not specified Other: Fluent in English Not pregnant or nursing

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: Not specified Endocrine therapy: Not specified Radiotherapy: Not specified Surgery: Not specified

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients determined to have recurrent, persistent, or progressive cancer and scheduled to undergo either oral or parenteral chemotherapy as prescribed by the treating physician.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 1999-11; Primary Completion 2002-11 (Actual); Study Completion 2002-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Calhoun, PhD, Study Chair — Robert H. Lurie Cancer Center
Locations (1):
- Robert H. Lurie Comprehensive Cancer Center, Northwestern University, Chicago, Illinois, United States